CLINICAL TRIAL: NCT00364026
Title: A Phase II Study to Evaluate the Effects of Darusentan on Safety and Efficacy in Subjects With Resistant Systolic Hypertension Receiving Combination Therapy With Three or More Antihypertensive Drugs, Including a Diuretic (Protocol DAR-201)
Brief Title: A Clinical Study to Evaluate the Effects of Darusentan on Safety and Efficacy in Subjects With Resistant Systolic Hypertension Receiving Combination Therapy With Three or More Blood Pressure Lowering Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol DAR-201
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2006-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — darusentan

INTERVENTIONS:
Drug: darusentan

SUMMARY:
This is a research study of a new experimental drug called darusentan. Darusentan is not currently approved by the U.S. Food and Drug Administration (FDA) for use in the United States, which means that a doctor cannot prescribe this drug. The purpose of this study is to determine if darusentan is effective in reducing systolic blood pressure in subjects with resistant systolic hypertension, despite treatment with full doses of three or more blood pressure lowering drugs, including a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are competent to provide written consent
* Aged 35 to 85 years
* Subjects with diabetes and/or chronic kidney disease must have a mean systolic blood pressure ≥130 mmHg
* All other subjects must have a mean systolic blood pressure ≥140 mmHg
* Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, including a diuretic
* Female subjects of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the time of Randomization.

Exclusion Criteria:

* Average sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg at Screening
* Serum ALT or AST >2X ULN
* Subjects who have experienced myocardial infarction, unstable angina, or a cerebrovascular accident (CVA) within 6 month of the Screening Visit; or sick sinus syndrome or second or third degree atrioventricular block, chronic atrial fibrillation or recurrent atrial tachyarrhythmia, recurrent ventricular tachycardia, or symptomatic bradycardia
* Implanted cardioverter defibrillator (ICD) that has fired for any arrhythmia within 3 months of Screening or implanted pacemakers
* Symptomatic CHF requiring treatment
* Hemodynamically significant valvular heart disease
* Hemodialysis or peritoneal dialysis; or history of renal transplant
* Diagnosis or recurrence of malignancy within the past 3 years
* Sleep apnea
* Subjects who perform alternating shift or night work
* Subjects who have participated in a clinical study involving another investigational drug or device within 1 month of the Screening Visit

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2005-07

PRIMARY OUTCOMES:
Co-primary efficacy measures are changes in trough sitting systolic BP from baseline through Weeks 8 and 10.

SECONDARY OUTCOMES:
Secondary efficacy measurements are change in trough sitting diastolic BP from baseline to study Week 10; change in mean 24-hour systolic BP, as measured by ABPM; and the percent of subjects who reached systolic BP goal after 10 weeks of treatment.